CLINICAL TRIAL: NCT04213599
Title: The Coronary Angiography Characteristic of Free Wall Ruptrue in ST-Elevation Myocardial Infarction Patients
Brief Title: The Angiography Characteristic of Free Wall Ruptrue in STEMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiamen Cardiovascular Hospital, Xiamen University (Other)
Responsible Party: Principal Investigator, Bin Wang, Ph D, Director, Xiamen Cardiovascular Hospital, Xiamen University
Other Study IDs: 9215443693
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: ST-Elevation Myocardial Infarction
Keywords: STEMI; Ruptrue; Angiography
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Anterior infarction: Patients with anterior ST-elevation myocardial infarction
  Interventions: Diagnostic Test: Coronary intervention
- Inferior infarction: Patients with inferior ST-elevation myocardial infarction
  Interventions: Diagnostic Test: Coronary intervention
- Lateral infarction: Patients with lateral ST-elevation myocardial infarction
  Interventions: Diagnostic Test: Coronary intervention

INTERVENTIONS:
Diagnostic Test: Coronary intervention — Patients with STEMI undergo coronary intervention

SUMMARY:
To analyze whether the location of myocardial infarction and infarct related artery are related to FWR.

DETAILED DESCRIPTION:
To know the characteristic of FWR that different location of STEMI and coronary distribution

ELIGIBILITY:
Inclusion Criteria:

1. Patients had to be ≥18 years of age, be admitted for STEMI
2. Accord with STEMI diagnostic criteria
3. STEMI patients anticipated to undergo angiography

Exclusion Criteria:

1. Pregnant
2. Acute stroke
3. Aortic dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STEMI patients anticipated to undergo angiography
Sampling Method: Non-Probability Sample
Enrollment: 14629 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of cardiac death | 30 days
  In-hospital cardiac death during 30 days
Number of free-wall rupture | 30 days
  The FWR after STEMI patients
Number of reperfusion arrhythmia | 30 days
  Reperfusion arrhythmia during coronary intervention

SECONDARY OUTCOMES:
FMC time | 30 days
  First Medical Contact time
Symptom onset to angiology time | 30 days
  The time from symptom onset to beginning of angiography

CONTACTS AND LOCATIONS:
Overall Officials: Bin Wang, PhD, Study Director — Xiamen Cardiovascular Hospital, Xiamen University
Locations (1):
- Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No